CLINICAL TRIAL: NCT04911504
Title: The Effects of Resilience and Self-efficacy on Nurses' Compassion Fatigue: A Cross-sectional Study
Brief Title: The Effects of Resilience and Self-efficacy on Nurses' Compassion Fatigue
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Jie Zhang, Principal investigator, Central South University
Other Study IDs: JZhang
Record Dates: First submitted 2021-05-27; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Compassion Fatigue; Self Efficacy; Resilience
Keywords: Compassion fatigue; Self-efficacy; Resilience; Nurses
MeSH Terms: conditions — Compassion Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire survey group: All nurses were recruited from 3 tertiary hospitals in central China from 3rd October, 2019 to 15th December, 2019. A total of 992 clinical nurses from different nursing departments were recruited through convenience sampling. Data were collected using General information questionnaire, the Professional Quality of Life Scale, the Connor-Davidson Resilience Scale and General Perceived Self-Efficacy Scale.

SUMMARY:
Among healthcare providers, nursing is a stressful and compassionate profession. Nurses empathetically support patients with pain, loneliness, disease and even confronted with death in line with their critically physical, mental, emotional, and spiritual needs and provide comfort, help, presence for them. Because nurses are frequently exposed to highly stressful and emotional situations, they suffer compassion fatigue (CF) over time under repeated exposures. CF will have a series of physiological, social, emotional, spiritual, and cognitive effects on nurses, threatening the existential integrity of them. The effects include high rates of anxiety and depressive disorders, decreased productivity, increased clinical errors, decreased quality of care and level of job satisfaction. Therefore, it is particularly important to pay attention to compassion fatigue to maintain mental health of nurses.

Compassion fatigue refers to that in the process of providing assistance, the helper bears the pain of the recipient due to empathy, which reduces the helper's own energy or interest.Based on a widespread conceptual model, CF consists of two constructs: burnout and secondary traumatic stress. Nurses are at a great risk of compassion fatigue. CF is gradually becoming a serious problem which can affect nurses' physical and psychological health, performance, job satisfaction and quality of care . Thus, investigating the prevalence of CF among nurses and its related factors are warranted to prevent CF among nursing population.

Research has studied the influencing factors of CF. Some studies have found that the demographic characteristics, worked related factors , the degree of exposure to traumatic events and psychological factors are important factors affecting nurses' compassion fatigue. Some studies suggest that resilience, social support, sense of control and meaningful recognition are negatively correlated with CF . Among them, resilience and self-efficacy are considered as important psychological factors affecting the individual's mental health, and they play an important role in the occurrence of CF.

The working pressure of clinical nurses comes from the situations that they are exposed to patients' traumatic events and give excessive empathy for a long-term. CF among nurses is an undesirable outcome caused by maladaptation to this pressure. What's more, resilience, and self-efficacy play an important role in individual coping and psychological adjustment in face of stressful events. Therefore, it is necessary to explore the roles of resilience and self-efficacy in the process of CF.

According to the theoretical path analysis of professional caregivers' quality of life, work environment, client environment and person environment factors have an influence on the development of compassion fatigue . Regarding to the psychological stress system , When confronted with stressful events, the individuals will have a stress response as a joint result of environmental factors and personnel factors. Thus, in accordance with the above two theories, being exposed to traumatic events is considered as a stressor, which could lead to CF. During this process, several external factors (work-related environmental factors) and internal factors (personality, social support) have effects on CF. In this study, resilience, and self-efficacy will be recognized as individual psychological characteristics and CF will be treated as a psychological change. Although there have been several studies on the predictors of CF in nurses around the world, limited knowledge exists in considering both internal factors (resilience and self-efficacy) and external predictive factors (demographic, work-related factors) of CF among nurses, especially in mainland China.

The study aims to investigate the level of compassion fatigue among Chinese nurses and test the influences of demographic characteristics, work-related factors, resilience, and self-efficacy on compassion fatigue.

DETAILED DESCRIPTION:
This study adopted a cross-sectional design. It was executed in accordance with STROBE Statement: guidelines for reporting observational studies.

Through convenience sampling, clinical nurses from different departments were recruited from three tertiary hospitals in central China.

According to the calculation method of the sample size regarding to the linear multiple regression, fixed model in G power software 3.1 was used. In this calculation, effect size f2=0.15, α= 0.05, 1-β=0.95, the study included 13 demographic variables, resilience and self-efficacy, 15 independent variables in total. The sample size calculated by G power software 3.1 is 199. Considering the 20% loss to follow-up rate and sampling error, the sample size was expanded to 239.

Measurement The general information questionnaire The social-demographic questionnaire was self-compiled and aimed to collect participants' demographic characteristics such as age, gender, educational level, marital status, working department, years of nursing experience, professional title, monthly income, shift work and physical conditions and so on.

Professional quality of life scale (Chinese version; ProQOL-CN) The Professional quality of life scale was used to evaluate the level of compassion fatigue. The original version was developed and then translated to Chinese. The scale has 30 items with three subscales including compassion satisfactory , burnout and secondary traumatic stress . Together, these latter two subscales measure compassion fatigue. A five-point Likert scale was used (1 = "never" to 5 = "very often") . A higher score of the compassion satisfaction subscale represents a higher level of compassion satisfaction, while a higher score of the burnout and secondary traumatic stress subscale indicates a higher risk of burnout and secondary traumatic stress. The score of each subscale lower than 22 represents a low level of compassion satisfaction, burnout, and secondary traumatic stress; score between 23 - 41 indicates an average level; and more than 42 suggests a high level . The Cronbach's alpha of the scale in this study was 0.722.

Connor-Davidson resilience scale (Chinese version; CD-RISC) The CD-RISC aimed to measure participants' resilience. The Chinese version of CD-RISC consists of three dimensions (tenacity, strength, and optimism) with 25 items. A five-point Likert scale was used (0 = "never" to 4 = "almost always"). The scale can effectively measure the resilience among clinical nurses and has good reliability and validity . The reliability of the CD-RISC among Chinese residents was 0.91 and the Cronbach's alpha of the scale in this study was 0.966.

General Perceived Self-Efficacy Scale (Chinese version; GSES) The GSES was used to measured participants' self-efficacy . The Chinese version consists of 10 items assessed by a four-point Likert scale (1=incorrect to 4=correct). The total scores range from 10 to 40, with higher total scores indicating higher levels of self-efficacy. The Cronbach's alpha of the scale in this study was 0.941.

Procedures Data were collected from 3rd October, 2019 to 15th December, 2019 and the data collection was completed by a researcher and two research assistants. First, the researchers informed the directors and head nurses from each hospital of the study's purpose and got their permission to recruit nurses. Then, researchers introduced the contents of the questionnaires to research assistants in the hospital and explained how to complete it. Lastly, researchers distributed a Wenjuanxing link (an online crowdsourcing platform in China) involved the electronic research questionnaires by scanning a Quick Response code to research assistants. According to the inclusion criteria, nurses who had interests could contact the researchers and research assistants in hospital to participate in the study. Wenjuanxing is a relatively secure platform and there is no risk of any data breach and leakage by a third-party.

ELIGIBILITY:
Inclusion Criteria:

* The hospital is a comprehensive hospital;
* Nurse have been registered and are on their duty;
* Nurses are currently engaged in clinical practice;
* Nurses are willing to participate in the study.

Exclusion Criteria:

* Nurses who are intern nurses or studying in other hospitals, or has been participated in other relevant studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the calculation method of the sample size regarding to the linear multiple regression, fixed model in G power software 3.1 was used. In this calculation, effect size f2=0.15, α= 0.05, 1-β=0.95, the study included 13 demographic variables, resilience and self-efficacy, 15 independent variables in total. The sample size calculated by G power software 3.1 is 199. Considering the 20% loss to follow-up rate and sampling error, the sample size was expanded to 239.
Sampling Method: Non-Probability Sample
Enrollment: 978 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
General information of participants questionnaire | baseline
  The general information of participants was measured by social-demographic questionnaire which was self-compiled and aimed to collect participants' demographic characteristics such as age, gender, educational level, marital status, working department, years of nursing experience, professional title, monthly income, shift work and physical conditions and so on.
Compassion fatigue of participants | baseline
  The Professional quality of life scale was used to evaluate the level of compassion fatigue. The original version was developed by Stamm and then translated to Chinese by Zheng, which was authorized by Stamm. The scale has 30 items with three subscales including compassion satisfactory , burnout and secondary traumatic stress. Together, these latter two subscales measure compassion fatigue. A five-point Likert scale was used (1 = "never" to 5 = "very often") . A higher score of the compassion satisfaction subscale represents a higher level of compassion satisfaction, while a higher score of the burnout and secondary traumatic stress subscale indicates a higher risk of burnout and secondary traumatic stress. The score of each subscale lower than 22 represents a low level of compassion satisfaction, burnout, and secondary traumatic stress; score between 23 - 41 indicates an average level; and more than 42 suggests a high level. The Cronbach's alpha of the scale in this study was 0.722.
Resilience of participants | baseline
  The Connor-Davidson resilience scale aimed to measure participants' resilience. The original version was developed by Connor and Davidson . Yu and Zhang translated it to Chinese after getting the authorization from the original developers. The Chinese version of CD-RISC consists of three dimensions (tenacity, strength, and optimism) with 25 items. A five-point Likert scale was used (0 = "never" to 4 = "almost always") . The scale can effectively measure the resilience among clinical nurses and has good reliability and validity. The reliability of the CD-RISC among Chinese residents was 0.91 and the Cronbach's alpha of the scale in this study was 0.966.
Self-Efficacy of participants | baseline
  The General Perceived Self-Efficacy scale developed by Scherbaum, was used to measured participants' self-efficacy. The Chinese version was translated by Wang . The scale consists of 10 items assessed by a four-point Likert scale (1=incorrect to 4=correct). The total scores range from 10 to 40, with higher total scores indicating higher levels of self-efficacy. The Cronbach's alpha of the scale in this study was 0.941.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya School of Nursing,Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The process of data collection cost a lot of human and material resources, some of the data was privacy information of participants, and so on.Considering this, it is improper to share these data.

REFERENCES:
- [Background] Ariapooran S. Compassion fatigue and burnout in Iranian nurses: The role of perceived social support. Iran J Nurs Midwifery Res. 2014 May;19(3):279-84. PMID 24949067
- [Background] Balinbin CBV, Balatbat KTR, Balayan ANB, Balcueva MIC, Balicat MGB, Balidoy TAS, Macindo JRB, Torres GCS. Occupational determinants of compassion satisfaction and compassion fatigue among Filipino registered nurses. J Clin Nurs. 2020 Mar;29(5-6):955-963. doi: 10.1111/jocn.15163. Epub 2020 Jan 13. PMID 31887244
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Background] Yao Y, Zhao S, Gao X, An Z, Wang S, Li H, Li Y, Gao L, Lu L, Dong Z. General self-efficacy modifies the effect of stress on burnout in nurses with different personality types. BMC Health Serv Res. 2018 Aug 29;18(1):667. doi: 10.1186/s12913-018-3478-y. PMID 30157926
- [Background] Zhang J, Zhang JP, Cheng QM, Huang FF, Li SW, Wang AN, Su P. The resilience status of empty-nest elderly in a community: A latent class analysis. Arch Gerontol Geriatr. 2017 Jan-Feb;68:161-167. doi: 10.1016/j.archger.2016.10.011. Epub 2016 Oct 26. PMID 27810664
- [Background] Sinclair S, Raffin-Bouchal S, Venturato L, Mijovic-Kondejewski J, Smith-MacDonald L. Compassion fatigue: A meta-narrative review of the healthcare literature. Int J Nurs Stud. 2017 Apr;69:9-24. doi: 10.1016/j.ijnurstu.2017.01.003. Epub 2017 Jan 12. PMID 28119163
- [Background] Zhang YY, Han WL, Qin W, Yin HX, Zhang CF, Kong C, Wang YL. Extent of compassion satisfaction, compassion fatigue and burnout in nursing: A meta-analysis. J Nurs Manag. 2018 Oct;26(7):810-819. doi: 10.1111/jonm.12589. Epub 2018 Aug 20. PMID 30129106
- [Result] Alharbi J, Jackson D, Usher K. Personal characteristics, coping strategies, and resilience impact on compassion fatigue in critical care nurses: A cross-sectional study. Nurs Health Sci. 2020 Mar;22(1):20-27. doi: 10.1111/nhs.12650. Epub 2019 Oct 31. PMID 31670474
- [Result] Arimon-Pages E, Torres-Puig-Gros J, Fernandez-Ortega P, Canela-Soler J. Emotional impact and compassion fatigue in oncology nurses: Results of a multicentre study. Eur J Oncol Nurs. 2019 Dec;43:101666. doi: 10.1016/j.ejon.2019.09.007. Epub 2019 Sep 12. PMID 31590071
- [Result] Cetrano G, Tedeschi F, Rabbi L, Gosetti G, Lora A, Lamonaca D, Manthorpe J, Amaddeo F. How are compassion fatigue, burnout, and compassion satisfaction affected by quality of working life? Findings from a survey of mental health staff in Italy. BMC Health Serv Res. 2017 Nov 21;17(1):755. doi: 10.1186/s12913-017-2726-x. PMID 29162095
- [Result] Guo YF, Luo YH, Lam L, Cross W, Plummer V, Zhang JP. Burnout and its association with resilience in nurses: A cross-sectional study. J Clin Nurs. 2018 Jan;27(1-2):441-449. doi: 10.1111/jocn.13952. Epub 2017 Sep 4. PMID 28677270
- [Result] Kelly L, Runge J, Spencer C. Predictors of Compassion Fatigue and Compassion Satisfaction in Acute Care Nurses. J Nurs Scholarsh. 2015 Nov;47(6):522-8. doi: 10.1111/jnu.12162. Epub 2015 Aug 19. PMID 26287741
- [Result] Nolte AG, Downing C, Temane A, Hastings-Tolsma M. Compassion fatigue in nurses: A metasynthesis. J Clin Nurs. 2017 Dec;26(23-24):4364-4378. doi: 10.1111/jocn.13766. Epub 2017 Apr 20. PMID 28231623
- [Result] Shen J, Yu H, Zhang Y, Jiang A. Professional quality of life: A cross-sectional survey among Chinese clinical nurses. Nurs Health Sci. 2015 Dec;17(4):507-15. doi: 10.1111/nhs.12228. Epub 2015 Aug 24. PMID 26303265
- [Result] Wang J, Okoli CTC, He H, Feng F, Li J, Zhuang L, Lin M. Factors associated with compassion satisfaction, burnout, and secondary traumatic stress among Chinese nurses in tertiary hospitals: A cross-sectional study. Int J Nurs Stud. 2020 Feb;102:103472. doi: 10.1016/j.ijnurstu.2019.103472. Epub 2019 Nov 13. PMID 31810017